CLINICAL TRIAL: NCT05591053
Title: Utility and Usability of ActivSight™ Laser Speckle Imaging in Visualization of Tissue Perfusion and Blood Flow During Esophageal Surgery in Humans
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Activ Surgical (Industry)
Collaborators: University of Pittsburgh Medical Center (Other); West Penn Allegheny Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ACF0052020
Record Dates: First submitted 2022-10-17; First posted 2022-10-24 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Esophagus Cancer; Esophageal Cancer; Esophageal Neoplasms; Esophageal Diseases; Esophageal Adenocarcinoma; Esophageal Squamous Cell Carcinoma; Esophagus SCC; Esophagus Tumor; Esophagus Adenocarcinoma; Esophagus Neoplasm
Keywords: laparoscopic; robot assisted surgery; gastrointestinal anastomoses; esophagectomy; esophageal surgery; thoracic surgery; alimentary surgery; perfusion; indocyanine green (ICG); laser speckle contrast imaging (LSCI); cancer; minimally invasive surgery (MIS)
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Diseases; Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma; Neoplasms

STUDY DESIGN:
Intervention Model Description: Target enrollment for the assessment of esophageal anastomoses is a total of 70 patients powered to detect ~ 2-3 cm discordance between ICG and LSCI lines of demarcation between well vascularized and less vascularized site in the gastric conduit. Since ActivSight™ can detect the difference of > 2 cm between perfused versus less perfused in comparison to ICG with 80 % confidence at p<0.05 in a sample size of n = 21, the investigators estimate that the study will require an accrual of 63 patients. With potential unforeseen dropout and mortality, the investigators recruit a total of 70 patients for the proposed study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- ActivSight Group (Experimental): Patients undergoing esophagectomy with ActivSight (n=70)
  Interventions: Device: ActivSight

INTERVENTIONS:
Device: ActivSight — Use of ActivSight in patients undergoing laparoscopic or robot assisted esophagectomy.

SUMMARY:
ActivSight™ combines an innovative form factor and proprietary software to deliver precise, objective, real-time visualization of blood flow and tissue perfusion intraoperatively for laparoscope-based surgery. A small adaptor that fits between any existing laparoscope and camera systems and a separate light source placed along any current commercial system will deliver objective real-time tissue perfusion and blood flow information intraoperatively.

Primary Objective: To determine the feasibility of ActivSight™ in detecting and displaying tissue perfusion and blood flow in the conduit and foregut anastomoses in esophageal resection/reconstructive surgery. The investigators will compare the precision and accuracy among the naked eye inspection, ICG and LSCI in assessing the vascularity of the conduit.

DETAILED DESCRIPTION:
Design:

* This is a prospective interventional cross-over study where ActivSight™ will be used in sequence to the standard practice of visualizing perfusion status of the conduit using the naked eye visual inspection and ICG during esophageal resection.
* Feasibility will be determined by technically successful completion of intended visualization.
* Safety will be determined through clinical assessments and evaluation of any adverse event.
* Assessment of preliminary efficacy will be performed through analysis of any intraoperative decisions made based on visual display as compared to standard endoscopic approach, or non-inferiority to ICG-based visualization and usability.
* Patient outcome and follow up to Postoperative day 28 will be monitored for clinical outcome.
* Target enrollment for the assessment of esophageal anastomoses is a total of seventy patients powered to detect ~ 2-3 cm discordance between ICG and LSCI lines of demarcation between well vascularized and less vascularized sites in the gastric conduit. Since ActivSight™ can detect the difference of > 2 cm between perfused versus less perfused in comparison to ICG with 80 % confidence at p<0.05 in a sample size of n = 21, the investigators estimate that the study will require an accrual of 63 patients. With potential unforeseen dropout and mortality, the investigators will recruit a total of 70 patients for the proposed study.

ELIGIBILITY:
INCLUSION CRITERIA

All patients age > 18 years old undergoing laparoscopic esophageal resection and reconstruction surgery; spoken command and literacy in the native language spoken at each participating center; ability to understand and follow study procedures; and having provided signed consent.

Diagnosis:

* All patients with a clinical suspicion and diagnosis of benign or malignant, small or large bowel lesions requiring surgical resection.
* Typical imaging as per standard workup findings including US, CT and/or MRI. Plain radiographs and contrast imaging may be obtained by referring physicians and are helpful for confirming the clinical diagnosis.

Location of pathology or resected segment:

* Target lesions can be located in any fore-, mid- or hindgut segments requiring reconstruction and anastomoses.

Prior therapy:

* Patients with prior surgery are eligible for enrollment.

Laboratory:

* Hemoglobin > 9 g/dL
* Platelet count ≥75,000/µL (may receive transfusions)
* Normal PT, PTT and INR < 1.5 x ULN (including patients on prophylactic anticoagulation)
* Renal function: Age-adjusted normal serum creatinine derived from Schwartz formula for estimating GFR by the CDC OR a creatinine clearance ≥60 mL/min/1.73 m2 for safe
* Adequate pulmonary function: Defined as no dyspnea at rest, and a pulse oximetry >94% on room air if there is clinical indication for determination.

EXCLUSION CRITERIA

* There is no exclusion criteria for ActivSightTM for esophageal surgery.
* Patients assigned to FDA cleared ICG-based visualization are contraindicated for any chronic renal dysfunction, potential drug interaction, history of allergy to ICG or anaphylaxis, known allergy to iodides, breast-feeding or being of reproductive age with pregnancy possible and not ruled out, and pregnancy.
* Patients currently in any investigational agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events in 28 days following use of ActivSight™ | 28 days
  To determine safety of ActivSight™ in patients undergoing esophageal surgery, as defined through clinical assessments and evaluation of use related adverse events intraoperatively and a routine follow up at 28 days following surgery. ActivSight™ will be deemed safe if no hardware (adaptor or light source)-related major (serious) adverse event is encountered in the treated patients and if less than 2 hardware-related minor adverse events are encountered.
  Adverse events will be summarized descriptively and tabulations on the type, severity, and relationship to application will be performed and any changes of outcomes from baseline on follow up will be examined using the nonparametric Wilcoxon rank test.
Preparation time of ActivSight™. | 1 day
  Rate on a scale of 1-5 (1 = Difficult to use or Unsatisfied - 5 = no training required or very satisfied): How easy was ActivSight to set up?
Latency of display of ActivSight™. | 1 day
  Rate on a scale of 1-5 (1 = Difficult to use or Unsatisfied - 5 = no training required or very satisfied): How specifically did ActivSight display the intended field and the target tissue of interest?
Resolution and objectivity of display of ActivSight™. | 1 day
  Rate on a scale of 1-5 (1 = Difficult to use or Unsatisfied - 5 = no training required or very satisfied): How was the display quality of ActivSight on the intended field and target tissue of interest?
Specificity of display of ActivSight™. | 1 day
  Specificity of display will serve as an outcome for feasibility. Yes/No question for surgeon: "Does the perfusion information displayed by ActivSightTM reflect the expected pattern of blood flow interruption?"
Usability of ActivSightTM by surgeon, as quantified by Likert scale. | 1 day
  Likert scale ratings will serve as an outcome for feasibility. Scale 1-5 question (1=strongly disagree, 2=slightly disagree, 3=neutral, 4=slightly agree, 5=strongly agree): "ActivSightTM was easy to use while operating."
Support personnel satisfaction with ActivSightTM, as quantified by Likert scale. | 1 day
  Likert scale ratings will serve as an outcome for feasibility. Scale 1-5 question (1=strongly disagree, 2=slightly disagree, 3=neutral, 4=slightly agree, 5=strongly agree): "ActivSightTM was easy to set up for the procedure."
User feedback on utility of relative perfusion unit display versus color heatmap | 1 day
  Likert scale ratings will serve as an outcome for feasibility. Scale 1-5 question (1=strongly disagree, 2=slightly disagree, 3=neutral, 4=slightly agree, 5=strongly agree):
Episodes of intraoperative decision change based on display | 1 day
  Yes/No if surgeons changed intraoperative planning/decisions based on ActivSight™, with additional details (what did they change and why) requested if yes.
Usability of the device by surgeon and support personnel satisfaction; | 1 day
  Likert scale ratings will serve as an outcome for feasibility. Scale 1-5 question (1=strongly disagree, 2=slightly disagree, 3=neutral, 4=slightly agree, 5=strongly agree):

SECONDARY OUTCOMES:
Ability of ActivSightTM to display perfusion. | 1 day
  ActivSightTM ability to display perfusion at a tissue level during gastrointestinal anastomoses is measured by the following Yes/No question for the surgeon: "Does ActivSightTM display tissue perfusion of the anatomy during anastomoses in comparison to ICG?"
Ability of ActivSightTM to display blood vessels. | 1 day
  ActivSightTM ability to display blood vessels during gastrointestinal anastomoses is measured by the following Yes/No question for the surgeon: "Does ActivSightTM display vascularity of the anatomy during anastomoses in comparison to ICG?"

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Pittsburgh Medical Center - Dept of Cardiothoracic Surgery, Pittsburgh, Pennsylvania
  - West Penn Hospital / Allegheny Health Network, Pittsburgh, Pennsylvania